CLINICAL TRIAL: NCT03464968
Title: A Randomized Phase II Study of mFOLFOX vs. mFOLFIRI in Advanced or Recurrent Biliary Tract Cancer Refractory to First Line Gemcitabine Plus Cisplatin
Brief Title: mFOLFOX vs. mFOLFIRI in Advanced or Recurrent Biliary Tract Cancer Refractory to First Line
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jin Won Kim, Clinical Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: biliary second line
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Biliary Cancer Metastatic
Keywords: second line; FOLFOX; FOLFIRI
MeSH Terms: interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOX (Experimental): D1 oxaliplatin 100mg/m2 over 2hr Leucovorin 100mg/m2 over 2hr 5FU 2400mg/m2 over 46hr Every 2 weeks
  Interventions: Drug: Oxaliplatin,5FU, leucovorin
- mFOLFIRI (Experimental): D1 Irinotecan 150mg/m2 over 2hr Leucovorin 100mg/m2 over 2hr 5FU 2400mg/m2 over 46hr Every 2 weeks
  Interventions: Drug: irinotecan,5FU, leucovorin

INTERVENTIONS:
Drug: Oxaliplatin,5FU, leucovorin — mFOLFOX
  Arms: mFOLFOX
Drug: irinotecan,5FU, leucovorin — mFOLFIRI
  Arms: mFOLFIRI

SUMMARY:
In second line with advanced or recurrent biliary tract cancer refractory to first line gemcitabine plus cisplatin, efficacy of mFOLFOX vs. mFOLFIRI will be evaluated at randomized phase 2 trial.

DETAILED DESCRIPTION:
1. brief enrollment criteria

   * histological confirmed
   * refractory to first line gemcitabine plus cisplatin
   * fit for chemotherapy
2. treatment arms A. mFOLFOX D1 oxaliplatin 100mg/m2 over 2hr Leucovorin 100mg/m2 over 2hr 5FU 2400mg/m2 over 46hr Every 2 weeks

   B. mFOLFIRI D1 Irinotecan 150mg/m2 over 2hr Leucovorin 100mg/m2 over 2hr 5FU 2400mg/m2 over 46hr Every 2 weeks
3. randomization - stratified by tumor site and performance status

ELIGIBILITY:
Inclusion Criteria:

* 20 years and older
* pathologically confirmed biliary tract cancer (adenocarcinoma) including intrahepatic, extrahepatic, gallbladder, ampulla of vater
* initially inoperable or recurrent
* ECOG 0-2
* as first line chemotherapy, refractory to gemcitabine/cisplatin (at least one cycle applied)
* evaluable or measurable lesion
* within 1 week, patients who meet below laboratory results (hemoglobin >9.0 g/dL, neutrophil >1000/uL, platelet> 75000/uL, serum creatinine < UNL * 1.5, AST/ALT < UNL*3, total bilirubin < UNL*1.5 (available for biliary drainage)
* patients who have ability to understand the purpose, benefit and harm for this trial, and the right to withdraw this trial in any time without any disadvantage

Exclusion Criteria:

* other cancer history
* pregnant or lactating
* uncontrolled medical condition such as infection or cardiovascular disease
* hypersensitivity to experimental drugs
* uncontrolled CNS metastasis, psychologic problem

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
6 months overall survival rate | 6months
  at 6 months from intervention treatment, overall survival rate

SECONDARY OUTCOMES:
response rate | 6months
  complete response, partial response
disease control rate | 6months
  complete response, partial response, stable disease
progression free survival | 6months
  from treatment start to progression or any cause of death
Number of Participants With Treatment-Related Adverse Events as Assessed by NCI CTC version 4.0 | 6months
  percentage of all patients

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi IS, Kim KH, Lee JH, Suh KJ, Kim JW, Park JH, Kim YJ, Kim JS, Kim JH, Kim JW. A randomised phase II study of oxaliplatin/5-FU (mFOLFOX) versus irinotecan/5-FU (mFOLFIRI) chemotherapy in locally advanced or metastatic biliary tract cancer refractory to first-line gemcitabine/cisplatin chemotherapy. Eur J Cancer. 2021 Sep;154:288-295. doi: 10.1016/j.ejca.2021.06.019. Epub 2021 Jul 22. PMID 34303267